CLINICAL TRIAL: NCT00420654
Title: Growth Hormone Treatment of Women With Turner Syndrome: Body Composition and Heart Function.
Brief Title: Growth Hormone Treatment of Women With Turner Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Britta E. Hjerrild (Other)
Responsible Party: Sponsor-Investigator, Britta E. Hjerrild, MD PhD Clinical assistent, University of Aarhus
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-BH-GH
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Turner Syndrome
Keywords: Turner syndrome; growth hormone treatment; positron emission tomography; heart
MeSH Terms: conditions — Turner Syndrome | interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A1 (Active Comparator)
  Interventions: Drug: Growth Hormone
- A2 (Placebo Comparator)
  Interventions: Drug: Placebo
- A3 (Other)
  Interventions: Other: Healthy controls

INTERVENTIONS:
Drug: Growth Hormone — 1.25 mg, 6 months
  Arms: A1
Drug: Placebo — Equivalent to 1.25 mg, 6 months
  Arms: A2
Other: Healthy controls — Healthy controls
  Arms: A3

SUMMARY:
Growth hormone treatment is used in girls with Turner syndrome to increase final height. The aim of this study is to evaluate the effect of growth hormone treatment on body composition and heart function in adult women with Turner syndrome. The hypothesis is that the fat mass will decrease and lean body mass will increase. There is only very limited documentation of the effect on the heart in this study population.

DETAILED DESCRIPTION:
This study is a randomised, double-blinded, controlled clinical trial to evaluate the effect of growth hormone (GH) treatment on adult women with Turner syndrome. The endpoints will be changes in body composition and heart function evaluated by echocardiography (ECHO) and positron emission tomography (PET).

Phase one: 6 months of GH or placebo treatment. Phase two: "open label" all participants are treated with GH for 12 months. At baseline, healthy controls will be examined, but will not receive any treatment

ELIGIBILITY:
Inclusion Criteria:

* Turner syndrome
* Age 20-40

Exclusion Criteria:

* Symptomatic heart disease
* Anti hypertensive treatment
* Untreated thyroid disease
* Adipositas (BMI > 35)
* Treatment with glucocorticoids
* Pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Body composition: fat mass and lean body mass | 6 months + 18 months
Myocardial perfusion and glucose uptake, evaluated by positron emission tomography | 6 months

SECONDARY OUTCOMES:
Heart function evaluated by echocardiography (conventional and tissue doppler) | 6 months + 18 months
Lipid profile | 6 months + 18 months
24 hour ambulatory blood pressure | 6 months + 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens S. Christiansen, prof. dr.med, Principal Investigator — University of Aarhus
Locations (1):
- Medical Department M (Endocrinology and Diabetes), Aarhus University Hospital, Aarhus, DK, Denmark